CLINICAL TRIAL: NCT07015450
Title: The Efficacy of Self-Manufactured 40% Dextrose Gel as Supplementary to Asymptomatic Transient Neonatal Hypoglycemia Treatment : A Randomized Controlled Trial
Brief Title: The Efficacy of Self-Manufactured 40% Dextrose Gel in Asymptomatic Transient Neonatal Hypoglycemia Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Budi Kemuliaan Hospital (Unknown); Universitas Indonesia, Cipto Mangunkusumo National General Hospital (Unknown); RS Prof. Dr. I.G.N.G Ngoerah (Unknown)
Responsible Party: Principal Investigator, Rosalina Dewi Roeslani, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KET-407/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Neonatal Hypoglycemia
Keywords: asymptomatic transient neonatal hypoglycemia; 40% dextrose gel
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Intervention group : given self manufactured 40% dextrose gel applied in buccal mucosa region plus standard therapy
  Interventions: Drug: self-manufactured 40% dextrose gel; Drug: Standard therapy
- Control Group (Placebo Comparator): Control group : given a standard therapy only
  Interventions: Drug: Standard therapy

INTERVENTIONS:
Drug: self-manufactured 40% dextrose gel — The self-manufactured 40% dextrose gel was applied in buccal mucosa region
  Arms: Intervention Group
Drug: Standard therapy — standard therapy for asymptomatic transient neonatal hypoglycemia

SUMMARY:
The goal of this clinical trial is to determine the efficacy of 40% dextrose gel therapy as an additional therapy for the management of asymptomatic transient neonatal hypoglycemia in high risk infants

The main question it aims to answer is:

Is 40% dextrose gel effective for the management of asymptomatic transient NH in high risk infants?

Researchers will compare the use of 40% dextrose gel as an additional therapy to the standard treatment and the use of breastmilk or formula milk according standard hypoglycemia treatment only to see if 40% dextrose gel is superior than standard therapy for management as asymptomatic transient NH in high risk infants.

Participants will :

* Receive 40% dextrose gel plus standard therapy or standard therapy only
* Blood glucose level measurement (30 minutes after intervention)

DETAILED DESCRIPTION:
Background: Neonatal hypoglycemia (NH) is a metabolic disorder that often occurs in the first few days of life. It is a potential cause of preventable brain injury and neonatal death. Most of hypoglycemia in high risk infants are transient and asymptomatic. One of the additional therapy for asymptomatic transient neonatal hypoglycemia is 40% dextrose gel. The 40% dextrose gel is a promising therapy because it is inexpensive, easy to administer and non-invasive.

Objective: To determine the efficacy of 40% dextrose gel therapy as an additional therapy for the management of asymptomatic transient NH in high risk infants.

Methods: A single-blind, randomized controlled trial was carried out in April-August 2023. The inclusion criteria were infants >34 weeks of gestational age and birth weight >1500 grams with blood sugar levels of 27-<47 mg/dL and without hypoglycemic symptoms. Block randomization was carried out in 60 eligible subjects. Subjects were allocated to 2 groups, the treatment group (40% dextrose gel plus standard therapy) and control group (standard therapy). The self-manufactured 40% dextrose gel was applied in buccal mucosa region. Blood glucose level was measured with glucometer 30 minutes after intervention. Data presented in descriptive and analyzed using chi-square and independent t-test with p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Infants with gestational age >34 weeks and birth weight >1500 grams with one of risk factors for hypoglycemia, such as baby with large for gestational age (LGA), small for gestational age (SGA), intrauterine growth restriction (IUGR), late preterm infants (LPIs), history of antenatal corticosteroid administration for 24 hours to 7 days before delivery; Maternal risk factors: hypertensive mothers, preeclampsia, diabetes type 1 or 2 mothers during or before pregnancy, consumed medication that caused hypoglycemia (terbutaline, b-blockers)
* Blood sugar levels at 0-4 hours after delivery are 27-<47 mg/dL,
* The parents agreed to participate in the research

Exclusion Criteria:

* birth asphyxia that require active resuscitation and neonatal intensive care unit (NICU) care
* infants with symptoms of hypoglycemia
* Infants who have absolute and relative contraindications for enteral and oral feeding.

Min Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Blood Glucose Serum Levels | From enrollment to 30 minutes after intervention
  Blood glucose level was measured from capillary blood with glucometer which validated every two weeks by supervised technician. Blood serum obtained by skilled health workers at 30 minutes after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Putu Mas Vina Paramitha Cempaka, Dr, Principal Investigator — Pediatric Subspecialist Consultant Program, Child Health Department, Faculty of Medicine - Universitas Indonesia, Cipto Mangunkusumo Hospital, Jakarta, Indonesia
Locations (3):
- Indonesia (3):
  - Prof IG.N.G Ngoerah General Hospital Denpasar, Denpasar, Bali
  - Budi Kemuliaan Hospital, Jakarta, Jakarta Special Capital Region
  - Child Health Department, Faculty of Medicine - Universitas Indonesia, Cipto Mangunkusumo Hospital, Jakarta, Indonesia, Jakarta, Jakarta, Jakarta, Jakarta Special Capital Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neonatal mortality - UNICEF DATA. Accessed October 30, 2023. https://data.unicef.org/topic/child-survival/neonatal-mortality/
- [Background] Edwards T, Harding JE. Clinical Aspects of Neonatal Hypoglycemia: A Mini Review. Front Pediatr. 2021 Jan 8;8:562251. doi: 10.3389/fped.2020.562251. eCollection 2020. PMID 33489995
- [Background] Vain NE, Chiarelli F. Neonatal Hypoglycaemia: A Never-Ending Story? Neonatology. 2021;118(5):522-529. doi: 10.1159/000514711. Epub 2021 Mar 22. PMID 33752207
- [Background] Committee on Fetus and Newborn; Adamkin DH. Postnatal glucose homeostasis in late-preterm and term infants. Pediatrics. 2011 Mar;127(3):575-9. doi: 10.1542/peds.2010-3851. Epub 2011 Feb 28. PMID 21357346
- [Background] Thornton PS, Stanley CA, De Leon DD, Harris D, Haymond MW, Hussain K, Levitsky LL, Murad MH, Rozance PJ, Simmons RA, Sperling MA, Weinstein DA, White NH, Wolfsdorf JI; Pediatric Endocrine Society. Recommendations from the Pediatric Endocrine Society for Evaluation and Management of Persistent Hypoglycemia in Neonates, Infants, and Children. J Pediatr. 2015 Aug;167(2):238-45. doi: 10.1016/j.jpeds.2015.03.057. Epub 2015 May 6. No abstract available. PMID 25957977
- [Background] Stanley CA, Rozance PJ, Thornton PS, De Leon DD, Harris D, Haymond MW, Hussain K, Levitsky LL, Murad MH, Simmons RA, Sperling MA, Weinstein DA, White NH, Wolfsdorf JI. Re-evaluating "transitional neonatal hypoglycemia": mechanism and implications for management. J Pediatr. 2015 Jun;166(6):1520-5.e1. doi: 10.1016/j.jpeds.2015.02.045. Epub 2015 Mar 25. No abstract available. PMID 25819173
- [Background] Hubbard EM, Hay WW Jr. The Term Newborn: Hypoglycemia. Clin Perinatol. 2021 Aug;48(3):665-679. doi: 10.1016/j.clp.2021.05.013. PMID 34353586
- [Background] Harris DL, Weston PJ, Harding JE. Incidence of neonatal hypoglycemia in babies identified as at risk. J Pediatr. 2012 Nov;161(5):787-91. doi: 10.1016/j.jpeds.2012.05.022. Epub 2012 Jun 23. PMID 22727868
- [Background] Alsaleem M, Saadeh L, Kamat D. Neonatal Hypoglycemia: A Review. Clin Pediatr (Phila). 2019 Nov;58(13):1381-1386. doi: 10.1177/0009922819875540. Epub 2019 Sep 26. No abstract available. PMID 31556318
- [Background] Thompson-Branch A, Havranek T. Neonatal Hypoglycemia. Pediatr Rev. 2017 Apr;38(4):147-157. doi: 10.1542/pir.2016-0063. PMID 28364046
- [Background] Adamkin DH. Neonatal hypoglycemia. Semin Fetal Neonatal Med. 2017 Feb;22(1):36-41. doi: 10.1016/j.siny.2016.08.007. Epub 2016 Sep 4. PMID 27605513
- [Background] Meneghin F, Manzalini M, Acunzo M, Daniele I, Bastrenta P, Castoldi F, Cavigioli F, Zuccotti GV, Lista G. Management of asymptomatic hypoglycemia with 40% oral dextrose gel in near term at-risk infants to reduce intensive care need and promote breastfeeding. Ital J Pediatr. 2021 Oct 9;47(1):201. doi: 10.1186/s13052-021-01149-7. PMID 34627324
- [Background] Sharma D, Shastri S, Sharma P. Intrauterine Growth Restriction: Antenatal and Postnatal Aspects. Clin Med Insights Pediatr. 2016 Jul 14;10:67-83. doi: 10.4137/CMPed.S40070. eCollection 2016. PMID 27441006
- [Background] Hu J, Benny P, Wang M, Ma Y, Lambertini L, Peter I, Xu Y, Lee MJ. Intrauterine Growth Restriction Is Associated with Unique Features of the Reproductive Microbiome. Reprod Sci. 2021 Mar;28(3):828-837. doi: 10.1007/s43032-020-00374-5. Epub 2020 Oct 26. PMID 33107014
- [Background] Samayam P, Ranganathan PK, Kotari UD, Balasundaram R. Study of Asymptomatic Hypoglycemia in Full Term Exclusively Breastfed Neonates in First 48 Hours of Life. J Clin Diagn Res. 2015 Sep;9(9):SC07-10. doi: 10.7860/JCDR/2015/14971.6610. Epub 2015 Sep 1. PMID 26500974
- [Background] Harris DL, Weston PJ, Signal M, Chase JG, Harding JE. Dextrose gel for neonatal hypoglycaemia (the Sugar Babies Study): a randomised, double-blind, placebo-controlled trial. Lancet. 2013 Dec 21;382(9910):2077-83. doi: 10.1016/S0140-6736(13)61645-1. Epub 2013 Sep 25. PMID 24075361
- [Background] Scheans P, Bennett C, Harris D. Using Dextrose (Glucose) Gel to Reverse Neonatal Hypoglycemia. Neonatal Netw. 2017 Jul 1;36(4):233-238. doi: 10.1891/0730-0832.36.4.233. PMID 28764827
- [Background] Makker K, Alissa R, Dudek C, Travers L, Smotherman C, Hudak ML. Glucose Gel in Infants at Risk for Transitional Neonatal Hypoglycemia. Am J Perinatol. 2018 Sep;35(11):1050-1056. doi: 10.1055/s-0038-1639338. Epub 2018 Mar 26. PMID 29579758
- [Background] Arimitsu T, Kasuga Y, Ikenoue S, Saisho Y, Hida M, Yoshino J, Itoh H, Tanaka M, Ochiai D. Risk factors of neonatal hypoglycemia in neonates born to mothers with gestational diabetes. Endocr J. 2023 May 29;70(5):511-517. doi: 10.1507/endocrj.EJ22-0521. Epub 2023 Mar 15. PMID 36792172
- [Background] Hawdon JM, Weddell A, Aynsley-Green A, Ward Platt MP. Hormonal and metabolic response to hypoglycaemia in small for gestational age infants. Arch Dis Child. 1993 Mar;68(3 Spec No):269-73. doi: 10.1136/adc.68.3_spec_no.269. PMID 8466261
- [Background] Barber RL, Ekin AE, Sivakumar P, Howard K, O'Sullivan TA. Glucose Gel as a Potential Alternative Treatment to Infant Formula for Neonatal Hypoglycaemia in Australia. Int J Environ Res Public Health. 2018 Apr 27;15(5):876. doi: 10.3390/ijerph15050876. PMID 29702618